CLINICAL TRIAL: NCT07168616
Title: Prospective Evaluation of Istanbul PSMA PET/CT Criteria for Selecting Candidates for Active Surveillance in Low-Risk Prostate Cancer
Brief Title: Study of PSMA PET/CT Imaging to Help Select Men With Low-Risk Prostate Cancer for Active Surveillance
Acronym: I-SELECT
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Yeditepe University (Other); Yedikule Training and Research Hospital (Other); Acibadem University (Other); Ankara Yildirim Beyazıt University (Other); University of Gaziantep (Other); Istanbul Training and Research Hospital (Other Government); Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Levent Kabasakal, Professor of Nuclear Medicine, Medical Doctor, Istanbul University - Cerrahpasa
Other Study IDs: 2024-KAEK-21/1153
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Low Risk Prostate Cancer; Clinically Significant Prostate Cancer
Keywords: PSMA PET/CT; Low risk prostate cancer; active surveillance; prostate cancer; clinically significant prostate cancer; Diagnosis of prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ga-68 PSMA11 PET/CT — delayed (120-minute) Ga-68 PSMA PET/CT and will be evaluated by using Istanbul PSMA PET/CT Criteria (IPPC)

SUMMARY:
This is a multicenter, prospective diagnostic accuracy study evaluating the Istanbul PSMA PET/CT Criteria (IPPC) for selecting patients with biopsy-confirmed low-risk prostate cancer (ISUP Grade 1) for active surveillance (AS). The study integrates delayed Ga-68 PSMA PET/CT imaging into the diagnostic pathway to refine patient stratification, minimize overtreatment and potentially reduce unnecessary biopsies and MRI, or exposing high-risk individuals to the danger of cancer progression if left untreated scans.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy in men and demonstrates heterogeneous clinical behavior. While many low-risk patients have indolent disease, a subset harbors clinically significant prostate cancer (csPCa) requiring early intervention. Active Surveillance (AS) is widely used to avoid overtreatment; however, current selection criteria-PSA, DRE, biopsy Gleason score, number of positive cores, PSA density, and mpMRI-lack sufficient predictive accuracy. Studies indicate that up to 30% of patients classified as low-risk by biopsy are found to have higher-grade disease at radical prostatectomy. The Istanbul PSMA PET/CT Criteria (IPPC) were developed by a multidisciplinary expert panel in Turkey to classify intraprostatic lesions on delayed (120-minute) Ga-68 PSMA PET/CT imaging into three risk categories:

* IPPC 1 No or homogeneous low uptake - safe for monitoring.
* IPPC 2: Indeterminate uptake - AS with close follow-up.
* IPPC 3: Focal, lentiform, high SUVmax ≥12 uptake in peripheral zone - definitive treatment recommended.

This study will evaluate the diagnostic performance of IPPC compared to standard mpMRI and biopsy findings, using radical prostatectomy pathology or long-term clinical follow-up as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* mpMRI performed within 3 months prior to enrollment
* Systematic or MRI-targeted prostate biopsy performed
* Biopsy-confirmed ISUP Grade 1 low-risk PCa
* Prostate biopsy report specifying tumor localization and number of positive cores
* Meets AS criteria: ISUP 1, PSA ≤10 ng/mL, PSAd >0.15 ng/mL², clinical stage cT1c-T2a, ≤3 positive cores
* Life expectancy ≥10 years
* No prior PSMA PET imaging
* No evidence of extra-prostatic disease on mpMRI
* Signed informed consent for study procedures

Exclusion Criteria:

* High-risk or unfavorable intermediate-risk PCa, or adverse histologies (neuroendocrine, ductal adenocarcinoma, basal cell carcinoma, TP53 or BRCA1/2 mutations if available)
* Prior prostate cancer treatment or prostate surgery
* MRI evidence of extracapsular extension, seminal vesicle invasion, or nodal metastasis
* History of pelvic radiotherapy
* Life expectancy <10 years
* Severe renal impairment
* Inability to comply with follow-up schedule

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only Turkish patients
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
1. Diagnostic Accuracy of the Istanbul PSMA PET/CT Criteria (IPPC) for Detecting Clinically Significant Prostate Cancer (csPCa) | Baseline imaging; confirmed at prostatectomy or through 2-year follow-up.
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the ROC curve (AUC) for IPPC classification in identifying csPCa, defined as ISUP Grade Group ≥2 on radical prostatectomy pathology or disease progression on long-term follow-up.

SECONDARY OUTCOMES:
Reduction in Repeat Biopsy Rate | Assessed over 2 years.
  Percentage of patients avoiding unnecessary repeat biopsies due to IPPC classification, compared with historical AS protocols

OTHER OUTCOMES:
Role of PSMA PET/CT During Active Surveillance | Baseline imaging; confirmed at prostatectomy or through 2-year follow-up.
  During follow-up, participants will undergo PSMA PET/CT either when clinical or biochemical progression is suspected, or annually even without evidence of progression. This will allow evaluation of whether PSMA PET/CT has a role in guiding patient management during Active Surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Kabasakal, Prof. MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (10):
- Turkey (Türkiye) (10):
  - Yeditepe University, Istanbul, Turkey
  - Bilkent Şehir Hastanesi, Ankara
  - Gazi Yaşargil Egitim ve Arastirma Hastanesi, Diyarbakır
  - Gaziantep Üniversitesi Şahinbey Araştırma ve Uygulama hastanesi, Gaziantep
  - Acibadem University Altunizade Hospital, Istanbul
  - Acibadem University Maslak Hospital, Istanbul
  - Haseki Eğitim ve Araştırma Hastanesi, Istanbul
  - Istanbul University-Cerrahpaşa, Istanbul
  - SBÜ Başakşehir Çam Sakura Şehir hastanesi, Istanbul
  - Sisli Hamidiye Etfal Eğitim ve Arastırma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seravalli J, Kumar M, Ragsdale SW. Rapid kinetic studies of acetyl-CoA synthesis: evidence supporting the catalytic intermediacy of a paramagnetic NiFeC species in the autotrophic Wood-Ljungdahl pathway. Biochemistry. 2002 Feb 12;41(6):1807-19. doi: 10.1021/bi011687i. PMID 11827525
- [Background] Drachenberg CB, Abruzzo LV, Klassen DK, Bartlett ST, Johnson LB, Kuo PC, Kumar D, Papadimitriou JC. Epstein-Barr virus-related posttransplantation lymphoproliferative disorder involving pancreas allografts: histological differential diagnosis from acute allograft rejection. Hum Pathol. 1998 Jun;29(6):569-77. doi: 10.1016/s0046-8177(98)80005-1. PMID 9635676
- [Background] Akcay K, Kibar A, Sahin OE, Demirbilek M, Beydagi G, Asa S, Aghazada F, Toklu T, Selcuk NA, Onal B, Kabasakal L. Prediction of clinically significant prostate cancer by [68 Ga]Ga-PSMA-11 PET/CT: a potential tool for selecting patients for active surveillance. Eur J Nucl Med Mol Imaging. 2024 Apr;51(5):1467-1475. doi: 10.1007/s00259-023-06556-y. Epub 2023 Dec 19. PMID 38112777
- [Background] Cornford P, van den Bergh RCN, Briers E, Van den Broeck T, Brunckhorst O, Darraugh J, Eberli D, De Meerleer G, De Santis M, Farolfi A, Gandaglia G, Gillessen S, Grivas N, Henry AM, Lardas M, van Leenders GJLH, Liew M, Linares Espinos E, Oldenburg J, van Oort IM, Oprea-Lager DE, Ploussard G, Roberts MJ, Rouviere O, Schoots IG, Schouten N, Smith EJ, Stranne J, Wiegel T, Willemse PM, Tilki D. EAU-EANM-ESTRO-ESUR-ISUP-SIOG Guidelines on Prostate Cancer-2024 Update. Part I: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2024 Aug;86(2):148-163. doi: 10.1016/j.eururo.2024.03.027. Epub 2024 Apr 13. PMID 38614820